CLINICAL TRIAL: NCT02971787
Title: Influence of Increased Salt Intake on Lactobacillus Abundance in Healthy Men
Brief Title: Salt Intake and Lactobacillus Abundance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Anja Maehler, Principle Investigator, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Tissue Salt 5
Record Dates: First submitted 2016-11-18; First posted 2016-11-23 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteers; Probiotics; Sodium
MeSH Terms: interventions — Probiotics; Salts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Probiotics and salt (Experimental): Lactobacillus enrichment and salt increase
  Interventions: Dietary Supplement: Probiotics; Dietary Supplement: Salt

INTERVENTIONS:
Dietary Supplement: Probiotics — Day 1-21: 2 capsules per day
  Other Names: Vivomixx
Dietary Supplement: Salt — Day 8-21: 10 tablets à 600 mg per day
  Other Names: Slow Sodium Tablets

SUMMARY:
To investigate the influence of an increased salt intake (6 g/d for 14 days) on the relative abundance of gut lactobillus species in healthy men

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* 18 - 50 years
* Body mass index 18,5 - 29,9 kg/m2

Exclusion Criteria:

* Clinically relevant heart, lung, liver, and kidney disease
* Current or chronic infections
* Habitual intake of probiotics or dietary supplements

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Decrease of relative abundance of four lactobacillus species | 14 days

SECONDARY OUTCOMES:
Increase of systolic blood pressure | 14 days
Increase of pulse wave velocity | 14 days
Increase of lymphocytic pro-inflammatory mediators | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Anja Maehler, PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Experimental and Clinical Research Center, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mahler A, Wilck N, Rauch G, Dechend R, Muller DN. Effect of a probiotic on blood pressure in grade 1 hypertension (HYPRO): protocol of a randomized controlled study. Trials. 2020 Dec 29;21(1):1032. doi: 10.1186/s13063-020-04973-0. PMID 33375942
- See also: Follow-up study — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-020-04973-0